CLINICAL TRIAL: NCT03727555
Title: Intrathecal and Intravenous Lentiviral Gene Therapy for X-linked Adrenoleukodystrophy (X-ALD)
Brief Title: IT and IV Lentiviral Gene Therapy for X-ALD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-18006
Record Dates: First submitted 2018-09-25; First posted 2018-11-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: X-linked Adrenoleukodystrophy
Keywords: X-linked adrenoleukodystrophy; Lentiviral vector; Intrathecal injection; Intravenous injection
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lentivirus-mediated delivery of ABCD1 to the CNS and the body (Experimental): Intrathecal and intravenous injections with lentiviral TYF-ABCD1 vector carrying the functional gene
  Interventions: Genetic: Intrathecal and intravenous LV gene therapy

INTERVENTIONS:
Genetic: Intrathecal and intravenous LV gene therapy — Direct IT and IV LV gene therapy to deliver high levels of LVs at 1-2×10^9 multiplicity of infection/ml which carry normal ABCD1 gene

SUMMARY:
This is a Phase I/II clinical trial of gene therapy for treating X-linked adrenoleukodystrophy using a high-safety, high-efficiency, self-inactivating lentiviral vector (LV) TYF-ABCD1 to functionally correct the defective gene. The objectives are to evaluate the safety and efficacy of the intrathecal and intravenous lentiviral gene transfer clinical protocol.

DETAILED DESCRIPTION:
X-linked adrenoleukodystrophy (X-ALD) is a devastating neurological disorder caused by mutations in the ABCD1 gene that encodes a peroxisomal ATP-binding cassette transporter (ABCD1). ABCD1 is responsible for transport of CoA-activated very long-chain fatty acids (VLCFA) into the peroxisome for degradation. X-ALD is clinically characterized with two main phenotypes: adrenomyeloneuropathy (AMN) and the inflammatory cerebral ALD. This disease presents most commonly in males. Approximately 50% of heterozygote females show some symptoms later in life. Approximately two-thirds of ALD patients will present with the childhood cerebral form of the disease, which is the most severe form. The disease is characterized by normal development in early childhood, followed by rapid degeneration to a vegetative state. ALD patients are normally treated with hematopoietic stem cell transplantation (HSCT) from a matched healthy donor. However, HSCT must be performed at a very early stage of the disease, which limits the therapeutic opportunities for juvenile or adult forms of ALD. This trial aims to treat ALD using a safety and efficiency improved self-inactivating lentiviral vector carrying a functional ABCD1 gene via intrathecal (IT) and intravenous (IV) injections to directly correct the genetic defect. This protocol targets not only early stage patients but also patients with symptoms. The direct LV injection approach aims to correct the pathologies associated with this genetic defect, and the IT and IV LV injections substantially simplify the treatment process, which reduces the risk associated with myeloablative chemotherapy during the HSCT treatment.

The objectives are to evaluate the safety of the advanced self-inactivating LV TYF-ABCD1, the direct in vivo gene transfer clinical protocol and the efficacy of the treatment, including assessment of vector distribution and the potential long-term correction of the ALD disease phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. X-ALD patients ≥ 1 year of age
2. ALD diagnosis of the brain: evaluation of the VLCFA value in plasma
3. Central imaging of the MRI to examine the damage on the CNS.
4. Neurological function score (NFS) ≥ 1
5. Parent / guardian / patient signing informed consent
6. Patients and their families have a strong willingness to participate in clinical trials, and are willing to bear all the consequences caused by the failure of the trial, and sign an informed consent form

Exclusion Criteria:

1. HIV positive patients
2. Stablized condition after statins, Lorenzo's oil, or diet to reduce VLCFA levels
3. Patients who are experiencing severe viral, bacterial or fungal infections, malignant tumors, heart abnormalities, liver dysfunction, or renal insufficiency
4. Cannot perform an MRI
5. Infection or dermatosis at pre-injection site

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of IT and IV injections of lentiviral TYF-ABCD1, determined by number of participants with treatment-related adverse events (AEs), according to scheduled assessments, vital signs, & physical examinations as assessed by CTCAE v4.0. | Minimum 1 day, maximum 1 year follow up
  Safety of direct IT and IV injections of lentiviral TYF-ABCD1, determined by number of participants with treatment-related adverse events (AEs), according to scheduled assessments, vital signs, & physical examinations as assessed by CTCAE v4.0. AEs & clinically significant abnormalities (meeting grade 3, 4, or 5 criteria according to CTCAE) will be summarized by maximum intensity & relationship to study drug(s). Grade 1 & 2 AEs will be summarized if related to study therapy.
Altered disease progression | Minimum 6 months, maximum 3 year follow up
  Altered disease progression based on biochemicaland neurological analysis.
Assess disease progression | Minimum 6 months, maximum 3 year follow up
  Assess disease progression based on MRI brain imaging analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No